CLINICAL TRIAL: NCT00073970
Title: A Trial Of COX-2 Inhibitors In PSA Recurrence After Definitive Radiation Or Radical Prostatectomy For Prostate Cancer
Brief Title: Celecoxib in Treating Patients With Relapsed Prostate Cancer Following Radiation Therapy or Radical Prostatectomy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study stopped due to increased cardiovascular risks associated with Celebrex
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LCCC 0109; UNC-01-SURG-655-ORC; CDR0000341468 (Other: PDQ number)
Record Dates: First submitted 2003-12-10; First posted 2003-12-11 (Estimated); Last update posted 2012-05-23 (Estimated); Status verified 2012-05

CONDITIONS: Prostate Cancer
Keywords: recurrent prostate cancer; stage I prostate cancer; stage II prostate cancer; adenocarcinoma of the prostate
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Celecoxib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: celecoxib — 400mg, given twice daily
  Other Names: Celebrex

SUMMARY:
RATIONALE: Celecoxib may stop the growth of cancer by stopping blood flow to the tumor and by blocking the enzymes necessary for tumor cell growth.

PURPOSE: Phase II trial to study the effectiveness of celecoxib in treating patients who have relapsed prostate cancer following radiation therapy or radical prostatectomy.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the effect of celecoxib on prostate-specific antigen (PSA) levels in patients with prostate cancer in biochemical relapse after prior definitive radiotherapy or radical prostatectomy.
* Compare the PSA doubling times in patients treated with this drug vs historical controls.
* Compare the PSA doubling times in patients treated with this drug vs pretreatment PSA values.
* Determine the time to clinical recurrence in patients treated with this drug.

OUTLINE: Patients receive oral celecoxib twice daily. Treatment continues for 5 years in the absence of disease progression. Patients may continue treatment beyond 5 years at the discretion of the treating physician.

PROJECTED ACCRUAL: A total of 100 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of clinically localized adenocarcinoma of the prostate

  * T1 or T2 disease
* Received prior primary treatment with definitive radiotherapy (at least 5,500 cGy) OR radical prostatectomy
* Biochemical relapse within 5 years after prior primary therapy, defined as 1 of the following:

  * Detectable and rising prostate-specific antigen (PSA) after surgery (at least 2 values above the residual cancer detection limit of the assay)
  * PSA at least 2 values above 1 ng/mL OR at least 3 rising values at any level after radiotherapy
* PSA no greater than 10 ng/mL

PATIENT CHARACTERISTICS:

Age

* Not specified

Performance status

* ECOG 0-2

Life expectancy

* Not specified

Hematopoietic

* Not specified

Hepatic

* ALT no greater than 2.5 times upper limit of normal

Renal

* Creatinine normal

Other

* No allergy to cyclooxygenase-2 inhibitors, aspirin, nonsteroidal anti-inflammatory drugs, or sulfa drugs
* No untreated peptic ulcer disease

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* No prior chemotherapy

Endocrine therapy

* More than 6 months since prior adjuvant or neoadjuvant hormonal therapy

  * Duration of prior adjuvant or neoadjuvant hormonal therapy must have been no more than 6 months

Radiotherapy

* See Disease Characteristics
* Prior salvage radiotherapy after prostatectomy allowed

Surgery

* See Disease Characteristics

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2003-04; Primary Completion 2005-06 (Actual); Study Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
Effect of COX-2 inhibitors on PSA level | 9 months
  To study the effect of COX-2 inhibitors on PSA level in patients who have only biochemical relapse after definitive radiation therapy or surgery for prostate cancer. In particular, to study the effect of celecoxib on PSA levels and PSA doubling times as compared to 1) historical controls (known and well-described median PSA doubling times of 9 months), and 2) pre-treatment PSA values and doubling times.

SECONDARY OUTCOMES:
Disease progression rate | 5 years
  Progression will be defined as evidence of biochemical relapse (increase in serum PSA levels on 3 successive determinations, provided that the increase is at least 5 ng/ml from baseline) or clinical objective progression or relapse - i.e. the development of new lesions by digital rectal exam (DRE) or enlargement of existing lesion, or the development of symptoms of clinical progression (specifically bony pain) which is confirmed by radiological imaging studies

CONTACTS AND LOCATIONS:
Overall Officials: Raj S. Pruthi, MD, Study Chair — UNC Lineberger Comprehensive Cancer Center
Locations (1):
- Lineberger Comprehensive Cancer Center at University of North Carolina - Chapel Hill, Chapel Hill, North Carolina, United States